CLINICAL TRIAL: NCT07012941
Title: An Application of Super-pulsed TFL vs Ho:YAG Laser in Retrograde Intrarenal Surgery for Upper Ureter and Renal Stones: A Multi-center Prospective Randomized Controlled Trial
Brief Title: Super-Pulsed Thulium Fiber Laser Versus Holmium:YAG Laser in Retrograde Intrarenal Surgery for Upper Ureteral and Renal Stones
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: RenJi Hospital (Other); Tongji Hospital (Other); West China Hospital (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Renmin Hospital of Wuhan University (Other); Beijing Friendship Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Beijing Tsinghua Changgeng Hospital (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Peking University Shenzhen Hospital (Other); Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Xu Kewei, Kewei Xu, MD, Ph.D, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SYSKY-2024-050-01
Record Dates: First submitted 2025-05-20; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Ureterolithiasis; Renal Calculi
Keywords: Super pulse thulium fiber laser (SPTFL); Ho:YAG laser; Lithotripsy; Ureteral Stone; Ureteroscopy; renal stone
MeSH Terms: conditions — Ureterolithiasis; Kidney Calculi; Nephrolithiasis | interventions — Ureteroscopy

STUDY DESIGN:
Intervention Model Description: Arm 1: Superpulse Thulium Fiber laser Arm 2: Holmium:YAG laser
Who Masked: Participant
Masking Description: Prior to the surgery, it is necessary to select the surgical technique and follow the trial protocol by opening an envelope in the specified sequence. This trial protocol follows a "single blind" format, meaning that the researcher is aware of the surgical method while the subject remains unaware.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superpulse Thulium Fiber laser (SPTFL) (Active Comparator): With the help of a Superpuled Thulium Fibre laser machine, the ureteral or renal stones that are going to be treated with the RIRS procedure are either fragmented or dusted as part of the procedure.
  Interventions: Device: Superpulse Thulium Fiber laser (SPTFL) ureteroscopy for treatment of upper urinary tract stone or renal stone
- Holmium: YAG laser (Active Comparator): With the help of a Holmium fibre laser machine, the ureteral or renal stones that are going to be treated with the RIRS procedure are either fragmented or dusted as part of the procedure.
  Interventions: Device: Holmium: YAG laser ureteroscopy for treatment of upper urinary tract stone or renal stone

INTERVENTIONS:
Device: Superpulse Thulium Fiber laser (SPTFL) ureteroscopy for treatment of upper urinary tract stone or renal stone — RIRS procedure for upper ureteral or renal stone lithotripsy with Superpulsed Thulium Laser
  Arms: Superpulse Thulium Fiber laser (SPTFL)
Device: Holmium: YAG laser ureteroscopy for treatment of upper urinary tract stone or renal stone — RIRS procedure for upper ureteral or renal stone lithotripsy with Holmium: YAG Laser
  Arms: Holmium: YAG laser

SUMMARY:
The holmium laser is currently considered the gold standard for lithotripsy on urinary lithiasis, whereas the super-pulsed thulium fibre laser is a relatively new technology. Through a multi-center prospective randomised clinical study that mainly aims to explore the effectiveness and safety of a super-pulsed fibre thulium laser compared to a holmium laser in the treatment of upper ureteral and renal stones (10mm<cumulative maximum diameter ≤ 25mm) in retrograde intrarenal surgery. The research participants are assigned randomly to undergo retrograde intrarenal surgery (RIRS) either using a super-pulsed thulium fibre laser or a holmium-YAG laser with an allocation ratio of 1:1. The secondary aim of this study is to provide high-level evidence for the development of diagnostic and treatment guidelines in the field of urolithiasis, both domestically and internationally. The outcomes of the RIRS procedures are compared for the two treatment arms.

DETAILED DESCRIPTION:
Endoscopic surgery is the predominant method for treating urinary tract stones. The field of surgery has progressed from traditional open procedures and percutaneous lithotripsy to more advanced techniques such as mini, micro, and ureteroscopy methods. RIRS, which stands for retrograde intrarenal surgery, is a therapeutic option for upper ureteric or renal stones that are less than 2cm. Although various energy systems have been employed for stone fragmentation during ureteroscopy, laser energy is the predominant method used for this purpose. Both domestic and foreign criteria recommend the holmium laser. The thermal effects of the Ho:YAG laser efficiently pulverise stones. As a result, it is currently the most widely used laser for conducting laser lithotripsy on stones in the urinary tract. Unfortunately, the holmium-YAG laser system has some intrinsic problems, such as different components having varying effects. 2. During the fragmentation process, the stone displacement is large and difficult to accurately control. 3. Some stones cannot be powdered, heat-damaged, or perforated. 4. Mucosal damage during fragmentation makes it easy to bleed and ooze. 5. The powdering efficiency is low, the fragmentation time is long, there is a lower energy conversion ratio, excessive heat generation in machines, noise, etc. Thus, clinical practice requires a new laser technology to overcome the holmium laser's limitations.

Thus, new laser systems are being created to fix the issue. The newest laser technology, super-pulsed thulium fiber laser (SPTFL), has promising results. A super-pulse fibre thulium laser is a pulsed fibre thulium laser that can be clinically used for lithotripsy. In 2005, in vitro experiments related to super-pulsed fibre thulium laser lithotripsy were first reported. Experimental data suggests that, compared with holmium laser, thulium laser has the following advantages in urinary tract stone lithotripsy: 1. TFL has higher lithotripsy efficiency, and the stone ablation speed is 1.5-4 times faster than that of Ho:YAG. 2. A safer lithotripsy with a 4-fold reduction in penetration depth and a limited temperature increase inside the cavity (up to 39 °C). 3. Lower costs: low maintenance costs, low fibre damage, low equipment volume (1/8), high energy conversion. Subsequently, an increasing number of in vitro experiments and clinical studies have been conducted internationally. However, there is a scarcity of studies in the literature that directly compare the effectiveness and stone free rates of the Holmium-YAG laser and SPTFL systems. Consequently, investigators are interested in conducting a formal multi-center prospective randomised clinical study to compare the two systems in RIRS.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤ Age ≤ 75 years old, regardless of gender, able to tolerate surgery;
2. Patients who have been confirmed by bilateral renal/urinary tract CT to have upper ureteral or renal stones, single or multiple, and are planning to undergo ureteroscopic lithotripsy for stone removal;
3. Confirmed by bilateral renal/urinary tract CT, the cumulative maximum diameter of stones is 10mm<cumulative maximum diameter ≤ 25mm;
4. Those who voluntarily participate and sign an informed consent form.

Exclusion Criteria:

1. Uncontrollable systemic hemorrhagic disease;
2. Severe spinal deformities, severe hip joint deformities, and difficulty in lithotomy position;
3. Uncontrolled urinary tract infections;
4. Any intracavitary surgery caused by anatomical factors of the urinary system cannot be performed;
5. Pregnant, planned pregnancy within 3 months, and lactating female patients;
6. The patients determined by the investigator to be unsuitable for this study include (but are not limited to): known to have human immunodeficiency virus (HIV) or AIDS; Suffering from mental illness; Infectious diseases;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Stone-Free Rate at 4 Weeks Postoperative (Percentage of Participants) | 4 week post-operative
  Urinary tract CT（Computed Tomography）scan at 4 weeks post-operative did not reveal residual stones or residual stones with a diameter ≤ 2 mm and no clinical symptoms were defined as stone clearance

SECONDARY OUTCOMES:
Intraoperative complication rate (Percentage of Participants) | During the procedure
  Includes ureteral or renal pelvis perforation, mucosal avulsion, ureteral rupture, conversion to other treatments, and success rate of ureteral access sheath insertion.
Change in Hemoglobin from Baseline (g/dL) | Within 24 hours postoperative
  Hemoglobin measured before and within 24 hours after surgery
Change in Serum Creatinine from Baseline (μmol/L) | Within 24 hours postoperative
  Serum creatinine measured before and within 24 hours after surgery
Change in Blood Urea Nitrogen from Baseline (mmol/L) | Within 24 hours postoperative
  BUN measured before and within 24 hours after surgery
Operative time (Minutes) | Decided immediately after the surgery
  Duration of operation
Lithotripsy time (Minutes) | intra-operation
  Time spent performing laser lithotripsy
Length of Hospital Stay (Days) | up to 30 days
  Total number of days the participant is hospitalized for the surgical procedure, from the day of surgery until discharge
Total hospitalization costs | Up to 3 months
  Total cost incurred during the participant's hospital stay for the surgical procedure, including all procedural and inpatient care charges
Postoperative Complications (Clavien-Dindo Classification, Percentage of Participants) | Up to 30 days post-operative
  Postoperative complications, Recording data according to the Clavien-Dindo classification such as infection, pain, ureteral stricture and other complications that result in the need for intervention or readmission or surgical revision following the RIRS procedure.
Number of Additional Staged Procedures (Count per Participant) | Up to 3 months post-operation
  Number of additional surgical procedures required due to incomplete stone clearance, based on imaging findings at the 4-week follow-up after the initial RIRS procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kewei Xu, MD, PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat sen Memorial Hospital of Sun Yat sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang W, Fan J, Huang G, Li J, Zhu X, Tian Y, Su L. Prevalence of kidney stones in mainland China: A systematic review. Sci Rep. 2017 Jan 31;7:41630. doi: 10.1038/srep41630. PMID 28139722
- [Background] Khan SR, Pearle MS, Robertson WG, Gambaro G, Canales BK, Doizi S, Traxer O, Tiselius HG. Kidney stones. Nat Rev Dis Primers. 2016 Feb 25;2:16008. doi: 10.1038/nrdp.2016.8. PMID 27188687
- [Background] Fried NM, Irby PB. Advances in laser technology and fibre-optic delivery systems in lithotripsy. Nat Rev Urol. 2018 Sep;15(9):563-573. doi: 10.1038/s41585-018-0035-8. PMID 29884804
- [Background] Teichmann HO, Herrmann TR, Bach T. Technical aspects of lasers in urology. World J Urol. 2007 Jun;25(3):221-5. doi: 10.1007/s00345-007-0184-5. Epub 2007 May 30. PMID 17534625
- [Background] Emiliani E, Kanashiro A, Angerri O. Lasers for stone lithotripsy: advantages/disadvantages of each laser source. Curr Opin Urol. 2023 Jul 1;33(4):302-307. doi: 10.1097/MOU.0000000000001092. Epub 2023 Mar 17. PMID 36927702
- [Background] Traxer O, Keller EX. Thulium fiber laser: the new player for kidney stone treatment? A comparison with Holmium:YAG laser. World J Urol. 2020 Aug;38(8):1883-1894. doi: 10.1007/s00345-019-02654-5. Epub 2019 Feb 6. PMID 30729311
- [Background] Hale GM, Querry MR. Optical Constants of Water in the 200-nm to 200-microm Wavelength Region. Appl Opt. 1973 Mar 1;12(3):555-63. doi: 10.1364/AO.12.000555. PMID 20125343
- [Background] Ventimiglia E, Doizi S, Kovalenko A, Andreeva V, Traxer O. Effect of temporal pulse shape on urinary stone phantom retropulsion rate and ablation efficiency using holmium:YAG and super-pulse thulium fibre lasers. BJU Int. 2020 Jul;126(1):159-167. doi: 10.1111/bju.15079. Epub 2020 May 18. PMID 32277557
- [Background] Solano C, Corrales M, Panthier F, Candela L, Doizi S, Traxer O. Navigating urolithiasis treatment: assessing the practicality and performance of thulium fiber laser, holmium YAG, and thulium YAG in real-world scenarios. World J Urol. 2023 Oct;41(10):2627-2636. doi: 10.1007/s00345-023-04487-9. Epub 2023 Jul 20. PMID 37468656
- [Background] Dorantes-Carrillo LA, Basulto-Martinez M, Suarez-Ibarrola R, Heinze A, Proietti S, Flores-Tapia JP, Esqueda-Mendoza A, Giusti G. Retrograde Intrarenal Surgery Versus Miniaturized Percutaneous Nephrolithotomy for Kidney Stones >1cm: A Systematic Review and Meta-analysis of Randomized Trials. Eur Urol Focus. 2022 Jan;8(1):259-270. doi: 10.1016/j.euf.2021.02.008. Epub 2021 Feb 21. PMID 33627307
- [Background] Jiao B, Luo Z, Xu X, Zhang M, Zhang G. Minimally invasive percutaneous nephrolithotomy versus retrograde intrarenal surgery in surgical management of upper urinary stones - A systematic review with meta-analysis. Int J Surg. 2019 Nov;71:1-11. doi: 10.1016/j.ijsu.2019.09.005. Epub 2019 Sep 12. PMID 31521837
- [Background] Li Z, Lai C, Shah AK, Xie W, Liu C, Huang L, Li K, Yu H, Xu K. Comparative analysis of retrograde intrarenal surgery and modified ultra-mini percutaneous nephrolithotomy in management of lower pole renal stones (1.5-3.5 cm). BMC Urol. 2020 Mar 16;20(1):27. doi: 10.1186/s12894-020-00586-6. PMID 32178654
- [Result] Martov AG, Ergakov DV, Guseynov M, Andronov AS, Plekhanova OA. Clinical Comparison of Super Pulse Thulium Fiber Laser and High-Power Holmium Laser for Ureteral Stone Management. J Endourol. 2021 Jun;35(6):795-800. doi: 10.1089/end.2020.0581. Epub 2021 Jan 13. PMID 33238763
- See also: A SKOLARIKOS,A NEISIUS,A PETRIK,et al.EAU Guidelines on Urolithiasis,2022 — http://uroweb.org/guideline/urolithiasis